CLINICAL TRIAL: NCT05980182
Title: SUCCEED: Engaging Black Men in Colorectal Cancer Screening (CRC) Screening
Brief Title: Engaging Black Men in Colorectal Cancer Screening
Acronym: SUCCEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MCC-21-18632; HM20023619 (Other: Virginia Commonwealth University); CA264067-01 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2023-07-27; First posted 2023-08-07 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer; CRC; Behavior
Keywords: Colorectal Screening behaviors
MeSH Terms: conditions — Colorectal Neoplasms; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailored Screen to Save (S2S) content (Experimental): Content to be delivered using a combination of short video and text-based information optimized for delivery via Quick Response (QR) codes for smartphones.
  Interventions: Behavioral: mHealth Application

INTERVENTIONS:
Behavioral: mHealth Application — Self-directed application (app) that is downloaded to the participant's personal device. The app contains five informational videos, that provide an orientation to the content on the app, and discuss what colorectal cancer is, and the type of CRC screening tests that are available as well as a video with a personal history. There is a a National Cancer Institute (NCI) risk calculation tool, and a family history infographic. Once the videos have been viewed participants have the option to indicate if they wish to receive a call from the healthcare clinic to discuss scheduling an appointment for screening.

SUMMARY:
To determine the unmet needs, attitudes, barriers and facilitators of African American (AA)/ Black men use of colorectal cancer screening and describe how community leaders such as barbers may act as Community Champions to educate and facilitate screening participation.

ELIGIBILITY:
Inclusion Criteria:

* Adult men
* Identify as Black or African American
* Work or live in Petersburg, VA or surrounding counties
* Eligible for colorectal cancer (CRC) screening at time of study enrollment

Exclusion Criteria:

* Inability to speak or read English
* Currently up-to-date with CRC screening

Ages: 45 Years to 74 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-05 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Thomson, Ph.D., Principal Investigator — Virginia Commonwealt University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Thomson MD, Shahab GH, Cooper-McGill CA, Sheppard VB, Hill SS, Preston M, Keen Ii L. Increasing Colorectal Cancer Screening Among Black Men in Virginia: Development of an mHealth Intervention. JMIR Form Res. 2024 Oct 10;8:e50028. doi: 10.2196/50028. PMID 39388688

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tailored Screen to Save (S2S) Content
Started | 30
Completed | 20
Not Completed | 10
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Arm/Group | Tailored Screen to Save (S2S) Content
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 30
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Colorectal Screening Status
Description: The number of participants that complete screening (any type)
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Screen to Save (S2S) Content
Number analyzed (Participants) | 30
Participants | 6

2. Secondary Outcome: Determine Feasibility of Mobile Health (mHealth) Application -Enrollment
Description: The number of men that enroll for the intervention (application)
Time Frame: Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Screen to Save (S2S) Content
Number analyzed (Participants) | 30
Participants | 30

3. Secondary Outcome: Determine the Feasibility of the mHealth Application-Videos
Description: The number of participants that view the videos
Time Frame: Week 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Screen to Save (S2S) Content
Number analyzed (Participants) | 30
Participants | 17

4. Secondary Outcome: Determine the Feasibility of the mHealth Application- Retention
Description: The number of participants that complete Questionnaires (>65%)
Time Frame: Baseline (Day 1), Week 2, and Week 12
Population: Number of participants that completed questionnaires during specified timepoints.
Measure: Number; unit: participants
Arm/Group | Tailored Screen to Save (S2S) Content
Number analyzed (Participants) | 30
participants
  Baseline Questionnaires | 28
  Week 2 Questionnaires | 10
  Week 12 Questionnaires | 20

5. Secondary Outcome: Determine the Feasibility of the mHealth Application- Clinic/ Screening Request
Description: The number of participants that respond to the request to contact clinic/ navigation services
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Screen to Save (S2S) Content
Number analyzed (Participants) | 30
Participants
  Responded Yes for contact | 7
  Responded No for contact | 21
  Did not Respond | 2

6. Secondary Outcome: Determine the Feasibility of the mHealth Application - Sharing Content
Description: The number of participants that share content on social network
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Tailored Screen to Save (S2S) Content
Number analyzed (Participants) | 30
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this trial.
Description: Adverse events were not collected for this trial.
Arm/Group | Tailored Screen to Save (S2S) Content
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT05980182/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT05980182/ICF_001.pdf